CLINICAL TRIAL: NCT04793321
Title: Impact of Baby Carrying Methods on Females Balance During Standing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamada Ahmed (Other)
Responsible Party: Sponsor-Investigator, Hamada Ahmed, Assistant Professor of Biomechanics, Faculty of Physical Therapy, Cairo University, Cairo University
Organization: Cairo University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: baby carrying methods
Record Dates: First submitted 2021-03-01; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2020-09

CONDITIONS: Balance; Distorted
Keywords: Biodex; baby caryying methods; Balance

STUDY DESIGN:
Intervention Model Description: A single group repeated measures design was used under which each participant had their balance tested during three conditions:
  1. holding nothing (unloaded).
  2. holding an infant mannequin in arms(arms).
  3. holding an infant mannequin in the baby carrier(carriers).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healty nulliparous females (Other): each participant did three conditions:
  1. holding nothing (unloaded).
  2. holding an infant mannequin in arms(arms).
  3. holding an infant mannequin in the baby carrier(carriers).
  Interventions: Device: Baby carrier; Device: Biodex Balance System; Other: Infant mannequin; Device: Biodex gait trainer 2 TM

INTERVENTIONS:
Device: Baby carrier — * It is made in china.
  * It is made of Cotton-Polyester.
  * It has 3 belts - 2 shoulder belts and one waist belt for superior lumbar support. Shoulder straps are padded and adjustable for the parent's comfort. It has webbing straps for shoulder and waist strap adjustment.
  * It is suitable for newborn to 12-months baby
  * It is available online at babyshopstores "https://www.babyshopstores.com/"
Device: Biodex Balance System — * The Biodex Balance System SD (The Biodex Balance System SD Model 945-300, 115 VAC, Shirley, NY, USA) is used to assess the balance in this study.
  * It is an objective device that measures dynamic postural stability. It uses a circular platform that allows up to 20˚of of platform tilt in a 360˚ range of motion.
  * The measures of postural stability score for BBS are the Overall Stability Index (OSI), Medial-Lateral Stability Index (MLSI), and Anterior-Posterior Stability Index (APSI). These indices are standard deviations that assess the path of sway around the zero point from the center of the platform and are measured in degrees. A high score in these stability indices indicates poor balance.
Other: Infant mannequin — The mannequin infant has 3 Kg which corresponds to the infant's age from birth until 1month. This weight is selected as it corresponds to the age at which the infants are frequently carried by the mother .
Device: Biodex gait trainer 2 TM — Gait Trainer 2™ ( model number:950-385, 115 VAC 50/60 Hz, made in the USA) is used for participants to walk on as walking is one of the most common daily life activities. because caregivers commonly walk while carrying their infants as it has a calming effect on crying infants
  It consists of :
  * Display: Use Audio and Visual Biofeedback - real-time biofeedback prompts patients into a proper gait pattern.
  * Heart Rate Monitoring
  * Handrail
  * Open Platform

SUMMARY:
The purpose of this study was to investigate the effect of different baby carrying methods (including carrying in arms and carrying in a baby carrier) in the females' balance during standing and walking.

DETAILED DESCRIPTION:
Babywearing is defined as using a supporting device that helps to keep an infant close to a caregiver's trunk.

The practice of babywearing has many benefits to both children and caregivers as it is an extension of "skin-to-skin care (SSC)" or "kangaroo care" which has well-known therapeutic benefits. Such benefits for the infant include: improve physical and cognitive state, good sleep, less likely to continuously cry, better breastfeeding, temperature stability.

For mothers, many benefits were found as well for example lower stress and anxiety levels, decrease in heart rate HR and blood pressure BP, higher breastfeeding rates, increase maternal satisfaction, increased bonding of mother with their neonate .

Despite the great advantage of infant carrying, there are many adverse effects on the musculoskeletal system and ergonomics of the mother. Women who carry their babies throughout the day will probably have similar consequences as carrying an extra load so pain and injuries will occur.

It has been reported that infant carrying in-arms caused acute muscle soreness in the ipsilateral upper limb that was used to support the infant over the left shoulder. While during the front infant carrying methods (ICMs), the pressure of the infant carrier shoulder straps caused shoulder discomfort and pain.

The front infant carrying position has the next highest fatigue score as it results in lower Metabolic equivalent (METS) and VO2max value which means that it places significant demand on the metabolic system.

It have been reported that the increased cost of carrying an infant in one's arms is the cause for the development of infant carrying tools rapidly.

Infant carrying is a form of exterogestation, just like in pregnancy, there is an alteration that swings the center of gravity of the body, shifts the postural balance, and increases the risk of falls .

Contrariwise, the usage of the carrier resulted in more similar postural control variables to the unloaded condition. Mannen and colleagues advised the use of babywearing as it provides a mechanical advantage to the caregiver.

Surprisingly, no study so far has quantified the actual balance changes with different carrying methods (including carrying in arms and carrying in a baby carrier) during typical movements of daily life, such as walking or standing upright.

Previous research has indicated that carrying externals loads elicits an increase in the center of pressure (COP) measures of postural sway during quiet standing .

Mathew W. Hill & Price reported that holding external loads during standing is an important issue for many daily and occupational activities and these external loads can affect postural stability, which is important for the mother's and fetus's safety. Also, holding a load in the hand may have restricted and/or delayed postural reactions.

From this perspective, both carrying methods are considered extra load and the question is that there any carrying methods that have an advantage over others concerning balance?

ELIGIBILITY:
Inclusion Criteria:

1. Had normal menstrual cycles.
2. All females were recruited on a day other than mese days.
3. Their age ranged from 20 to 35 years old.
4. Their body mass index ranged from 18-30 kg/m².
5. Had no experience with babywearing or in arm-carrying methods

Exclusion Criteria:

* Subjects were excluded if they had the following criteria:

  1. Females who had irregular menstrual cycles.
  2. Females who used oral contraceptive drugs or hormonal supplementary and injections through the previous 3 months.
  3. Females who had Musculoskeletal disorders or pain in the upper and lower extremities in the prior 6 months.
  4. Females complained of knee, ankle, or back pain.
  5. Females with a severe chronic illness that interfere with balance such as vestibular dysfunction.
  6. Any health condition that could interfere with the ability to maintain balance was excluded.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2021-02-17 (Actual)

PRIMARY OUTCOMES:
APSI | 20 second
  Anterior-Posterior Stability Index
MLSI | 20 second
  Medial-Lateral Stability Index
OSI | 20 second
  the Overall Stability Index

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Amel Mohamed Yousef, Professor, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy/ Cairo University, Giza, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Inanir A, Cakmak B, Hisim Y, Demirturk F. Evaluation of postural equilibrium and fall risk during pregnancy. Gait Posture. 2014 Apr;39(4):1122-5. doi: 10.1016/j.gaitpost.2014.01.013. Epub 2014 Feb 2. PMID 24630464
- [Background] Brown MB, Digby-Bowl CJ, Todd SD. Assessing Infant Carriage Systems: Ground Reaction Force Implications for Gait of the Caregiver. Hum Factors. 2018 Mar;60(2):160-171. doi: 10.1177/0018720817744661. Epub 2017 Dec 15. PMID 29244534